CLINICAL TRIAL: NCT00804063
Title: Serum Citrate in Diagnosis and Follow-up for Glaucoma
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Sponsor
Other Study IDs: EK 325/08
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Glaucoma
Keywords: glaucoma; citrate
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, serum, aqueous
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: glaucoma patients
  Interventions: Procedure: drawing blood sample
- 2: non-glaucoma controls
  Interventions: Procedure: drawing blood sample

INTERVENTIONS:
Procedure: drawing blood sample — fasting blood sample

SUMMARY:
Glaucoma might be a mitochondria associated disease. Since citrate is a major component in mitochondrial metabolism its determination in blood might serve as a biomarker.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* glaucoma

Exclusion Criteria:

* Active ocular inflammation
* Ocular Hypertension
* Nephropathy
* Alcohol-, Drug abuse
* Mitochondriopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary university center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
serum citrate level | 1

SECONDARY OUTCOMES:
urine citrate | 1

CONTACTS AND LOCATIONS:
Overall Officials: David Goldblum, MD, Principal Investigator — University Hospital, Basel, Switzerland; Josef Flammer, MD, Study Chair — University Hospital, Basel, Switzerland; Selim Orguel, MD, Study Director — University Hospital, Basel, Switzerland; Stephan Fraenkl, MD, Principal Investigator — University Hospital, Basel, Switzerland; Fabrizio Branca, MD, Principal Investigator — University Basel
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland